CLINICAL TRIAL: NCT00620061
Title: A Multi-center, Open-labeled Study of the Long-term Safety and Efficacy of Lubiprostone in Patients With Opioid-induced Bowel Dysfunction
Brief Title: Opioid-induced Bowel Dysfunction: Long-Term Assessment of Lubiprostone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBD06S1
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2018-03

CONDITIONS: Opioid-Induced Bowel Dysfunction
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Experimental): Lubiprostone: 24 mcg capsule twice daily (BID) for 36 weeks
  Interventions: Drug: Lubiprostone 24

INTERVENTIONS:
Drug: Lubiprostone 24 — 24 mcg capsules for oral administration
  Other Names: Amitiza

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of lubiprostone administration in participants with opioid-induced bowel dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Has completed 12 weeks of blinded treatment in NCT00595946 or NCT00597428
* Will continue to be treated consistently for chronic, non-cancer-related pain with any full agonist opiate and will continue opiate therapy for the duration of the study
* Willing to continue to abstain from use of disallowed medications as defined per protocol

Exclusion Criteria:

* Has newly diagnosed impaired renal function identified at the Screening Visit [i.e., serum creatinine concentration > 1.8 milligrams per deciliter (mg/dL)]
* Has experienced an unexplained and/or clinically significant weight loss defined as > 5% within 90 days prior to Screening Visit.
* Has plans to participate in another trial with an investigational drug or device during the course of the extension study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (123):
- United States (120):
  - The Birmingham Pain Center, Birmingham, Alabama
  - Simon Williamson Clinic, PC, Hueytown, Alabama
  - Alabama Orthopedic Clinic, Mobile, Alabama
  - Clinical Research Advantage, Inc./ Mesa Family Medical Center, Mesa, Arizona
  - Redpoint Research, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Clinical Research Advantage, Inc., Phoenix, Arizona
  - Clinical Research Advantage, Inc. / East Valley Family Physicians, PLC, Tempe, Arizona
  - Clinical Research Advantage, Inc., Tempe, Arizona
  - Premiere Pharamaceutical Research, LLC, Tempe, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Verona Clinical Research, Inc., Tucson, Arizona
  - Advanced Clinical Therapeutics, LLC, Tucson, Arizona
  - Paradigm Clinical Research, Inc., Tucson, Arizona
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - Wilson and Charani, Tucson, Arizona
  - Arkansas Pain Research, Hot Springs, Arkansas
  - Teton Research, LLC, Little Rock, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - Orange County Clinical Trials, Anaheim, California
  - Advanced Pain Institute, Arcadia, California
  - Impact Clinical Trials, Beverly Hills, California
  - Digestive and Liver Disease Specialists, Garden Grove, California
  - RX Clinical Research, Inc., Garden Grove, California
  - Loma Linda University, Loma Linda, California
  - Pasadena Rehabilitation Institute, Pasadena, California
  - Northern California Research Corporation, Sacramento, California
  - Rider Research Group, San Francisco, California
  - ShahShreenath Clinical Service, Yorba Linda, California
  - Clinicos, LLC, Colorado Springs, Colorado
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Advanced Diagnostic Pain Treatment Center, New Haven, Connecticut
  - Meridien Research, Brooksville, Florida
  - Century Clinical Research Inc, Daytona Beach, Florida
  - International Medical Research, Daytona Beach, Florida
  - Clinical Physiology Associates/Clinical Study Center, Fort Myers, Florida
  - Southeastern Integrated Medical, PL dba Florida, Gainesville, Florida
  - Century Clinical Research, Holly Hill, Florida
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Drug Study Institute, Jupiter, Florida
  - Sunrise Medical Research, Inc., Lauderdale Lakes, Florida
  - Kenneth W. Ponder, MD, PA, Niceville, Florida
  - North Miami Research Inc., North Miami, Florida
  - DMI Health Care Group, Inc., Pinellas Park, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Meridien Research, St. Petersburg, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Pinnacle Trials Inc., Atlanta, Georgia
  - North Georgia Premier Research, Dawsonville, Georgia
  - Best Clinical Research, Decatur, Georgia
  - Drug Studies America, Marietta, Georgia
  - Millenium Pain Center, Bloomington, Illinois
  - University of Illinois at Chicago: Department of Medicine, Chicago, Illinois
  - Apex Medical Research, AMR, Inc, Chicago, Illinois
  - Redhead Research Inc., Peoria, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Davis Clinic, PC, Indianapolis, Indiana
  - Intergrated Clinical Trial Services, Inc, West Des Moines, Iowa
  - The Pain Treatment Center of the Bluegrass, Lexington, Kentucky
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - The Willis-Knighton Interventional Pain Center, Shreveport, Louisiana
  - Pain and Rehabilitation Medicine, Bethesda, Maryland
  - Columbia Medical Practice/ RxTrials, Inc., Columbia, Maryland
  - Brigham and Women's Hosptial, Chestnut Hill, Massachusetts
  - MedVadis Research Corporation, Wellesley Hills, Massachusetts
  - Center for Clinical Studies, Dearborn, Michigan
  - Apex Medical Research, AMR, Inc., Flint, Michigan
  - Professional Clinical Research - Interlochen, Interlochen, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - Medical Research Associates, Traverse City, Michigan
  - Center for Digestive Health, Troy, Michigan
  - MAPS Applied Research Center, Edina, Minnesota
  - Medex Healthcare Research Inc., St Louis, Missouri
  - Montana Neuroscience Institute Foundation / Montana Spine and Pain Center, Missoula, Montana
  - Office of Stephen H. Miller, MD, Las Vegas, Nevada
  - Affiliated Clinical Research, Inc., Las Vegas, Nevada
  - Ladder Family Practice, Las Vegas, Nevada
  - Impact Clinical Trials, Las Vegas, Nevada
  - Gastroenterology Research Associates, LLC, Cedar Knolls, New Jersey
  - Central Jersey Medical Research Center, Elizabeth, New Jersey
  - Virtua Lumberton Family Physicians, Lumberton, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - NYU Pain Management Center, New York, New York
  - Research Across America, New York, New York
  - University of Rochester, Pain Treatment Center, Rochester, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Duke University Medical Center, Durham, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Glenway Family Medicine, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - RAS Health Ltd., Marion, Ohio
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - McBride Clinic, Oklahoma City, Oklahoma
  - Memorial Clinical Research, Oklahoma City, Oklahoma
  - Pain Research of Oregon, LLC, Eugene, Oregon
  - Medford Medical Clinic, LLP, Medford, Oregon
  - Affinity Research, Portland, Oregon
  - Lehigh Gastroenterology Associates, Allentown, Pennsylvania
  - Albert Einstein Healthcare Network Einstein Pain Institute, Philadelphia, Pennsylvania
  - Jeffry A. Lindenbaum DO, PC, Yardley, Pennsylvania
  - Trident Institute of Medical Research, LLC, North Charleston, South Carolina
  - Southeastern Clinical Research, Chattanooga, Tennessee
  - Comprehensive Pain Specialists, PLLC, Hendersonville, Tennessee
  - Integrity Clinical Research, LLC, Milan, Tennessee
  - Texas Familicare Clinical Research, Hurst, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Advanced Research Institute, Ogden, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Hampton Roads Institution for Performance and Sports Medicine, Portsmouth, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Northwest Gastroenterology Associates, Bellevue, Washington
  - VAMC Milwaukee, Milwaukee, Wisconsin
- Canada (3):
  - Health Sciences Centre Pain Clinic, Winnipeg, Manitoba
  - AIM Health Group London North, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 4 December 2007 to 29 September 2009 at 137 recruitment sites in the United States (n=134) and Canada (n=3)
Groups:
- Lubiprostone: Lubiprostone: 24 mcg capsules twice daily (BID) for 36 weeks
Period: Overall Study
Arm/Group | Lubiprostone
Started | 439
Completed | 286
Not Completed | 153

BASELINE CHARACTERISTICS:
Arm/Group | Lubiprostone
Number analyzed (Participants) | 439
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263
  Male | 176
Region of Enrollment [Number; unit: participants]
  United States | 436
  Canada | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Weekly Spontaneous Bowel Movements (SBMs) Per Month
Description: A Spontaneous Bowel Movement (SBM) is defined as any bowel movement (BM) that did not occur within the 24-hour period following use of a rescue medication.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Intent-to-treat population with evaluable SBM data during the given month
Measure: Mean (Standard Deviation); unit: Weekly SBMs
Groups:
- All Participants: Lubiprostone: 24 mcg capsules twice daily (BID)
Arm/Group | All Participants
Number analyzed (Participants) | 439
Weekly SBMs
  Baseline | 1.4 (0.98)
  Month 1: number analyzed (Participants) | 420
  Month 1 | 4.9 (2.72)
  Month 2: number analyzed (Participants) | 406
  Month 2 | 4.9 (2.62)
  Month 3: number analyzed (Participants) | 374
  Month 3 | 5.0 (2.76)
  Month 4: number analyzed (Participants) | 348
  Month 4 | 5.0 (2.71)
  Month 5: number analyzed (Participants) | 330
  Month 5 | 5.0 (2.82)
  Month 6: number analyzed (Participants) | 312
  Month 6 | 5.0 (2.86)
  Month 7: number analyzed (Participants) | 301
  Month 7 | 5.1 (2.93)
  Month 8: number analyzed (Participants) | 279
  Month 8 | 5.3 (2.91)
  Month 9: number analyzed (Participants) | 260
  Month 9 | 5.2 (3.19)

2. Primary Outcome: Mean Weekly Bowel Movements (BMs) Per Month
Description: A Bowel Movement (BM) is defined as any BM (whether spontaneous or not)
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Intent-to-treat population with evaluable BM data during the given month
Measure: Mean (Standard Deviation); unit: Weekly BMs
Arm/Group | All Participants
Number analyzed (Participants) | 439
Weekly BMs
  Baseline: number analyzed (Participants) | 224
  Baseline | 2.4 (1.38)
  Month 1: number analyzed (Participants) | 423
  Month 1 | 5.0 (2.73)
  Month 2: number analyzed (Participants) | 410
  Month 2 | 5.0 (2.63)
  Month 3: number analyzed (Participants) | 378
  Month 3 | 5.2 (2.70)
  Month 4: number analyzed (Participants) | 349
  Month 4 | 5.1 (2.67)
  Month 5: number analyzed (Participants) | 332
  Month 5 | 5.1 (2.79)
  Month 6: number analyzed (Participants) | 314
  Month 6 | 5.1 (2.85)
  Month 7: number analyzed (Participants) | 302
  Month 7 | 5.2 (2.90)
  Month 8: number analyzed (Participants) | 283
  Month 8 | 5.4 (2.88)
  Month 9: number analyzed (Participants) | 262
  Month 9 | 5.3 (3.15)

3. Secondary Outcome: Number of Participants Classified as Monthly Responders
Description: A weekly SBM frequency rate is calculated as (168 x Number of SBMs / Number of hours observed).
  A participant with an SBM frequency rate between 3 and 4 was considered a moderate responder. A subject with an SBM frequency rate higher than 4 was considered a full responder. If a subject was a moderate responder or full responder for at least half the weeks in a month, then he or she was considered a monthly responder.
Time Frame: Months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Lubiprostone: 24 mcg capsules twice daily (BID) for 9 months
Arm/Group | All Participants
Number analyzed (Participants) | 439
Participants
  Month 1 | 322
  Month 2 | 323
  Month 3 | 291
  Month 4 | 270
  Month 5 | 259
  Month 6 | 250
  Month 7 | 239
  Month 8 | 233
  Month 9 | 202

4. Secondary Outcome: Straining Associated With Spontaneous Bowel Movements by Month
Description: Participants rate the straining associated with the SBM on a scale where 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe The highest score is 4, and lower scores are better.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Intent-to-treat with evaluable data at the given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 439
score on a scale
  Baseline: number analyzed (Participants) | 383
  Baseline | 2.7 (0.87)
  Month 1: number analyzed (Participants) | 426
  Month 1 | 1.7 (0.85)
  Month 2: number analyzed (Participants) | 412
  Month 2 | 1.7 (0.85)
  Month 3: number analyzed (Participants) | 384
  Month 3 | 1.6 (0.84)
  Month 4: number analyzed (Participants) | 362
  Month 4 | 1.7 (0.83)
  Month 5: number analyzed (Participants) | 345
  Month 5 | 1.6 (0.85)
  Month 6: number analyzed (Participants) | 325
  Month 6 | 1.7 (0.84)
  Month 7: number analyzed (Participants) | 314
  Month 7 | 1.7 (0.86)
  Month 8: number analyzed (Participants) | 295
  Month 8 | 1.6 (0.87)
  Month 9: number analyzed (Participants) | 281
  Month 9 | 1.6 (0.92)

5. Secondary Outcome: Stool Consistency of Spontaneous Bowel Movements by Month
Description: Participants rate each spontaneous bowel movement on a scale where 0 = very loose, 1 = loose, 2 = normal, 3 = hard, 4 = very hard (little balls) The highest score is 4, but the best score is 2.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Intent-to-treat with evaluable data at the given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 439
score on a scale
  Baseline: number analyzed (Participants) | 383
  Baseline | 3.0 (0.84)
  Month 1: number analyzed (Participants) | 426
  Month 1 | 2.3 (0.75)
  Month 2: number analyzed (Participants) | 412
  Month 2 | 2.2 (0.73)
  Month 3: number analyzed (Participants) | 384
  Month 3 | 2.2 (0.74)
  Month 4: number analyzed (Participants) | 362
  Month 4 | 2.2 (0.72)
  Month 5: number analyzed (Participants) | 345
  Month 5 | 2.2 (0.70)
  Month 6: number analyzed (Participants) | 325
  Month 6 | 2.2 (0.68)
  Month 7: number analyzed (Participants) | 314
  Month 7 | 2.2 (0.70)
  Month 8: number analyzed (Participants) | 295
  Month 8 | 2.2 (0.66)
  Month 9: number analyzed (Participants) | 281
  Month 9 | 2.2 (0.70)

6. Secondary Outcome: Constipation Severity by Month
Description: Participants rate the severity of their constipation on a scale where 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.
  The highest score is 4, but the best score is 0.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Intent-to-treat with evaluable scores at the given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 439
score on a scale
  Baseline | 2.4 (0.72)
  Month 1: number analyzed (Participants) | 426
  Month 1 | 1.5 (0.93)
  Month 2: number analyzed (Participants) | 417
  Month 2 | 1.5 (0.94)
  Month 3: number analyzed (Participants) | 386
  Month 3 | 1.5 (0.93)
  Month 4: number analyzed (Participants) | 363
  Month 4 | 1.5 (0.96)
  Month 5: number analyzed (Participants) | 344
  Month 5 | 1.4 (0.95)
  Month 6: number analyzed (Participants) | 325
  Month 6 | 1.4 (0.94)
  Month 7: number analyzed (Participants) | 314
  Month 7 | 1.4 (0.94)
  Month 8: number analyzed (Participants) | 298
  Month 8 | 1.4 (0.97)
  Month 9: number analyzed (Participants) | 279
  Month 9 | 1.4 (0.99)

7. Secondary Outcome: Abdominal Bloating by Month
Description: Participants rate their bloating on a scale where 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.
  The highest score is 4, but the best score is 0.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Intent-to-treat with evaluable data at the given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 439
score on a scale
  Baseline | 2.2 (0.74)
  Month 1: number analyzed (Participants) | 426
  Month 1 | 1.6 (0.88)
  Month 2: number analyzed (Participants) | 417
  Month 2 | 1.5 (0.90)
  Month 3: number analyzed (Participants) | 386
  Month 3 | 1.5 (0.91)
  Month 4: number analyzed (Participants) | 363
  Month 4 | 1.5 (0.90)
  Month 5: number analyzed (Participants) | 344
  Month 5 | 1.5 (0.92)
  Month 6: number analyzed (Participants) | 325
  Month 6 | 1.5 (0.91)
  Month 7: number analyzed (Participants) | 314
  Month 7 | 1.5 (0.93)
  Month 8: number analyzed (Participants) | 298
  Month 8 | 1.5 (0.95)
  Month 9: number analyzed (Participants) | 278
  Month 9 | 1.5 (0.95)

8. Secondary Outcome: Abdominal Discomfort by Month
Description: Participants rate their abdominal discomfort on a scale where 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.
  The highest score is 4, but the best score is 0.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Intent-to-treat with evaluable data at the given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 439
score on a scale
  Baseline | 2.2 (0.67)
  Month 1: number analyzed (Participants) | 426
  Month 1 | 1.5 (0.82)
  Month 2: number analyzed (Participants) | 417
  Month 2 | 1.4 (0.82)
  Month 3: number analyzed (Participants) | 386
  Month 3 | 1.4 (0.84)
  Month 4: number analyzed (Participants) | 363
  Month 4 | 1.4 (0.83)
  Month 5: number analyzed (Participants) | 344
  Month 5 | 1.4 (0.86)
  Month 6: number analyzed (Participants) | 325
  Month 6 | 1.4 (0.85)
  Month 7: number analyzed (Participants) | 314
  Month 7 | 1.4 (0.85)
  Month 8: number analyzed (Participants) | 298
  Month 8 | 1.4 (0.89)
  Month 9: number analyzed (Participants) | 279
  Month 9 | 1.4 (0.91)

9. Secondary Outcome: Bowel Habit Regularity by Month
Description: Participants rate their bowel habit regularity on a balanced scale of 1 to 7 where 1=Very Regular and 7=Very Irregular.
  The highest score is 7, but the best score is 1.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Intent-to-treat with evaluable data at the given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 439
score on a scale
  Baseline | 4.7 (1.59)
  Month 1: number analyzed (Participants) | 426
  Month 1 | 3.6 (1.39)
  Month 2: number analyzed (Participants) | 415
  Month 2 | 3.6 (1.38)
  Month 3: number analyzed (Participants) | 386
  Month 3 | 3.5 (1.42)
  Month 4: number analyzed (Participants) | 363
  Month 4 | 3.5 (1.45)
  Month 5: number analyzed (Participants) | 344
  Month 5 | 3.5 (1.47)
  Month 6: number analyzed (Participants) | 324
  Month 6 | 3.5 (1.50)
  Month 7: number analyzed (Participants) | 314
  Month 7 | 3.5 (1.47)
  Month 8: number analyzed (Participants) | 298
  Month 8 | 3.4 (1.49)
  Month 9: number analyzed (Participants) | 279
  Month 9 | 3.4 (1.51)

10. Secondary Outcome: Treatment Effectiveness by Month
Description: Participants rate treatment effectiveness on a scale where 0 = not at all effective, 1 = a little bit effective, 2 = moderately effective, 3 = quite a bit effective, 4 = extremely effective.
  The highest and best score is 4.
Time Frame: Months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Intent-to-treat with evaluable data at the given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 439
score on a scale
  Month 1: number analyzed (Participants) | 426
  Month 1 | 2.1 (0.98)
  Month 2: number analyzed (Participants) | 415
  Month 2 | 2.1 (1.02)
  Month 3: number analyzed (Participants) | 386
  Month 3 | 2.2 (1.04)
  Month 4: number analyzed (Participants) | 363
  Month 4 | 2.2 (1.05)
  Month 5: number analyzed (Participants) | 344
  Month 5 | 2.2 (1.05)
  Month 6: number analyzed (Participants) | 324
  Month 6 | 2.2 (1.04)
  Month 7: number analyzed (Participants) | 314
  Month 7 | 2.3 (1.05)
  Month 8: number analyzed (Participants) | 298
  Month 8 | 2.3 (1.08)
  Month 9: number analyzed (Participants) | 279
  Month 9 | 2.3 (1.09)

11. Secondary Outcome: Mean Weekly Complete SBMs by Month
Description: Participants rate each SBM as complete if their bowels feel completely empty after the SBM
Time Frame: Months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Intent-to-treat with evaluable data at the time point
Measure: Mean (Standard Deviation); unit: Weekly Complete SBMs
Arm/Group | All Participants
Number analyzed (Participants) | 439
Weekly Complete SBMs
  Month 1: number analyzed (Participants) | 348
  Month 1 | 3.1 (2.26)
  Month 2: number analyzed (Participants) | 335
  Month 2 | 3.4 (2.27)
  Month 3: number analyzed (Participants) | 317
  Month 3 | 3.6 (2.47)
  Month 4: number analyzed (Participants) | 280
  Month 4 | 3.6 (2.40)
  Month 5: number analyzed (Participants) | 273
  Month 5 | 3.7 (2.64)
  Month 6: number analyzed (Participants) | 255
  Month 6 | 3.7 (2.62)
  Month 7: number analyzed (Participants) | 239
  Month 7 | 3.9 (2.79)
  Month 8: number analyzed (Participants) | 231
  Month 8 | 3.9 (2.69)
  Month 9: number analyzed (Participants) | 199
  Month 9 | 4.2 (2.95)

12. Secondary Outcome: Mean Weekly Complete BMs by Month
Description: Participants rate each BM as complete if their bowels feel completely empty after the BM
Time Frame: Months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Intent-to-treat with evaluable data at the time point
Measure: Mean (Standard Deviation); unit: Weekly Complete BMs
Arm/Group | All Participants
Number analyzed (Participants) | 439
Weekly Complete BMs
  Month 1: number analyzed (Participants) | 350
  Month 1 | 3.1 (2.26)
  Month 2: number analyzed (Participants) | 342
  Month 2 | 3.4 (2.28)
  Month 3: number analyzed (Participants) | 321
  Month 3 | 3.6 (2.46)
  Month 4: number analyzed (Participants) | 285
  Month 4 | 3.7 (2.38)
  Month 5: number analyzed (Participants) | 274
  Month 5 | 3.8 (2.65)
  Month 6: number analyzed (Participants) | 258
  Month 6 | 3.8 (2.62)
  Month 7: number analyzed (Participants) | 243
  Month 7 | 3.8 (2.78)
  Month 8: number analyzed (Participants) | 236
  Month 8 | 3.9 (2.69)
  Month 9: number analyzed (Participants) | 206
  Month 9 | 4.1 (2.96)

ADVERSE EVENTS:
Time Frame: 9 months plus 7 days for follow-up
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 1/439
Serious Adverse Events (participants affected / at risk) | 34/439
Other Adverse Events (participants affected / at risk) | 100/439
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=439)
Gastroenteritis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Papilloma Viral Infection (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Nocardiosis (Infections and infestations) | 1
Meningitis Aseptic (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Abscess Limb (Infections and infestations) | 1
Septic Shock (Infections and infestations) | 1
Abdominal Abcess (Infections and infestations) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Coranary Artery Disease (Cardiac disorders) | 2
Myocardial Infarction (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Pain (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Oesophageal Mass (Gastrointestinal disorders) | 1
Abdominal Adhesions (Gastrointestinal disorders) | 1
Mental Status Changes (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Cognitive Disorder (Nervous system disorders) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1
Multiple Fractures (Injury, poisoning and procedural complications) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Jugular Vein Thrombosis (Vascular disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Cavitation (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=439)
Nausea (Gastrointestinal disorders) | 39
Diarrhoea (Gastrointestinal disorders) | 42
Upper Respiratory Tract Infection (Infections and infestations) | 28
Back Pain (Musculoskeletal and connective tissue disorders) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days